CLINICAL TRIAL: NCT03655522
Title: NAVX-010 - A Phase I, Double-Blind, Placebo-Controlled, Single-Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Subjects
Brief Title: NAVX-010-Phase I Tolerability and Pharmacokinetic Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Algenis SpA (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CLN 14-030
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Safety

STUDY DESIGN:
Intervention Model Description: This was a double-blind, placebo-controlled, randomized, single ascending dose, sequential group study. Each subject participated in only 1 treatment period.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAVX-010 (Active Comparator): Dose levels of NAVX-010 were 2, 8, 25, 50, and 75 mcg. Doses were administered as IM injections into the deltoid muscle in the fasted state. The IMP was supplied in glass vials containing 1.2 mL solution at a total GTX 2 and GTX 3 concentration of 42 mcg/mL (at a relative epimer ratio of 62% GTX 2:38% GTX 3).
  Interventions: Drug: NAVX-010
- Placebo (Placebo Comparator): Placebo was of identical appearance to the IMP, and was administered into the deltoid muscle in the fasted state.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAVX-010 — Dose levels of NAVX-010 were 2, 8, 25, 50, and 75 mcg. Four patients per active group. Each subject participated in only 1 treatment period.
  Other Names: Gonyautoxin 2/3
  Arms: NAVX-010
Drug: Placebo — There were two Placebos per group.
  Other Names: Placebo of NAVX-010
  Arms: Placebo

SUMMARY:
This was a double-blind, placebo-controlled, randomized, single ascending dose, sequential group study. Each subject participated in only 1 treatment period.

The primary objective was to determine the safety of single intramuscular (IM) injections of NAVX 010 in healthy subjects. The secondary objective was to determine the single dose pharmacokinetics (PK) of Gonyautoxin 2 (GTX 2) and Gonyautoxin 3 (GTX 3) following IM administration of NAVX 010 in healthy subjects.

Thirty subjects were studied in 5 groups (Groups A to E); each group consisted of 6 subjects, of which 4 subjects received the Investigational Medicinal Product and 2 subjects received placebo. All subjects completed the study and data for all subjects were included in the safety analyses. A total of 20 subjects received NAVX-010 and were included in the PK population and subsequent PK analysis.

DETAILED DESCRIPTION:
This was a double-blind, placebo-controlled, randomized, single ascending dose, sequential group study. Each subject participated in only 1 treatment period.

The primary objective was to determine the safety of single intramuscular (IM) injections of NAVX-010 in healthy subjects. The secondary objective was to determine the single dose pharmacokinetics (PK) of Gonyautoxin 2 (GTX 2) and Gonyautoxin 3 (GTX 3) following IM administration of NAVX-010 in healthy subjects.

Thirty subjects were studied in 5 groups (Groups A to E); each group consisted of 6 subjects, of which 4 subjects received the Investigational Medicinal Product (IMP; NAVX-010) and 2 subjects received placebo. All subjects completed the study and data for all subjects were included in the safety analyses. A total of 20 subjects received NAVX-010 and were included in the PK population and subsequent PK analysis.

This study comprised healthy male subjects of any ethnic origin, aged between 18 and 45 years, inclusive, and with a body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.

Dose levels of NAVX-010 were 2, 8, 25, 50, and 75 mcg. Doses were administered as IM injections into the deltoid muscle in the fasted state. The IMP was supplied in glass vials containing 1.2 mL solution at a total GTX 2 and GTX 3 concentration of 42 mcg/mL (at a relative epimer ratio of 62% GTX 2:38% GTX 3).

Placebo was of identical appearance to the IMP, and was administered into the deltoid muscle in the fasted state.

Single IM injections were administered in each group. Blood and urine samples were collected for the analysis of plasma and urinary concentrations of GTX 2 and GTX 3, and the following PK parameters for GTX 2 and GTX 3 were calculated: area under the concentration-time curve (AUC) from time 0 up to the time of last quantifiable plasma concentration (AUC0 t), AUC from time 0 to 24 hours postdose (AUC0-24), AUC from time 0 extrapolated to infinity (AUC0 ∞), percentage of AUC that is due to extrapolation from the time of last quantifiable concentration to infinity (%AUCextrap), maximum observed plasma concentration (Cmax), time of the maximum observed plasma concentration (tmax), time of last quantifiable plasma concentration (tlast), time before the start of absorption (tlag), apparent plasma terminal elimination half life (t½), apparent total plasma clearance (CL/F), apparent volume of distribution during the terminal elimination phase (Vz/F), amount of drug excreted in urine (Ae), percentage of dose excreted in urine (Fe), and renal clearance (CLR).

Safety evaluations included adverse events (AEs), vital signs, 12 lead electrocardiogram (ECG), telemetry, clinical laboratory evaluations, physical examination, and clinical study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* males
* between 18 and 45 years of age
* body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive
* body weight between 50 kg and 100 kg inclusive
* Subjects must be in good health, as determined by:
* medical history
* physical examination (at check-in)
* vital sign assessment
* 12-lead ECG
* clinical laboratory evaluations
* Subjects must be able to understand and respond to the clinical study questionnaire
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

* Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception (such as a condom with spermicidal oam/gel/film/cream/suppository), or to refrain from donating sperm from the time of dosing until 3 months after study drug administration.
* Male subjects whose partners are of child-bearing potential must also agree to use an additional highly effective method of contraception.
* Subjects who have donated;
* blood or platelets in the 3 months prior to screening
* plasma in the 7 days prior to screening
* Subjects who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator or consume alcohol within 48 hours prior to the screening visit and prior to check-in.
* Subjects who have smoked more than 10 cigarettes per day or the equivalent in tobacco use (e.g. chewing tobacco, eCigarettes and smoking cessation products [nicotine patch or gum]) during the 3 months prior to screening.
* Subjects who have used the following within 7 days prior to study drug administration, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety:
* any over-the-counter systemic or topical medication
* herbal remedies
* vitamin supplements
* mineral supplements
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days prior to study drug administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Subjects who have received:
* any prescribed systemic or topical medication within 15 days prior to study drug administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* slow release medicinal formulations considered to still be active within 15 days prior to study drug administration, unless in the opinion of the Investigator, the medication will not interfere with the study procedures or compromise safety.
* coumarins (e.g. warfarin) at any time in the subject's lifetime.
* Subjects who have an abnormality in heart rate, blood pressure, temperature, oxygen saturation or respiration rate that, in the opinion of the Investigator, increases the risk of participating in the study, at screening and prior to study drug administration.
* Specific exclusion criteria at screening and/or prior to dosing are heart rate <40 bpm or >110 bpm, systolic blood pressure <90 mmHg or >150 mmHg, diastolic blood pressure <40 mmHg or >90 mmHg, oxygen saturation <94%, confirmed by a repeat assessment.
* Subjects with a positive urine drug or alcohol screen at screening or first admission.
* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study, at screening and prior to study drug administration.
* Specific exclusion criterion at screening and/or prior to dosing is QTcF value >450 ms, confirmed by a repeat assessment.
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have been administered an investigational drug (new chemical entity) in the 30 days prior to study drug administration.
* Subjects with a significant history of drug allergy as determined by the Investigator, including known or suspected allergy to any of the study drug components.
* Subjects with a known or suspected shellfish allergy or a positive skin prick test for shellfish allergy at screening or first admission.
* Subjects who have any clinically significant abnormal physical examination finding at check-in (Day -1 or Day -2). Specific exclusion criterion is any skin condition or finding that would limit a local injection site examination.
* Subjects who have any clinically significant allergic condition (excluding non-active hayfever) as determined by the Investigator.
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders as determined by the Investigator.
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
* Subjects who have any clinically significant abnormal laboratory safety findings, in the opinion of the Investigator (one repeat assessment is acceptable), at screening and prior to study drug administration.
* Specific exclusion criteria at screening and/or prior to dosing are fasting serum glucose <60 mg/dL or >115 mg/dL, serum phosphorous >1.5 х upper limit of normal (ULN), serum blood urea nitrogen >1.5 х ULN, serum alanine aminotransferase (ALT) >1.5 х ULN, serum aspartate aminotransferase (AST) >1.5 х ULN, serum total bilirubin >1.5 х ULN, serum creatinine >1.5 х ULN, hemoglobin <12 g/100 mL.
* Subjects who:
* are known to have serum hepatitis
* are carriers of the hepatitis B surface antigen (HBsAg)
* are carriers of the hepatitis C antibody
* have a positive result to the test for human immunodeficiency virus (HIV) antibodies.
* Subjects who have previously received a dose in this study.
* Subjects who, in the opinion of the Investigator, should not participate in the study.
* Subjects with a history of complications with anesthesia, such as malignant hyperthermia.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2015-09-02 (Actual)

PRIMARY OUTCOMES:
Adverse events related to NAVX-010 | Monitored from dosing day until 5 days after dosed
  Any signs or symptoms will be observed and elicited at least once a day by open questioning. Subjects will also be encouraged to spontaneously report AEs occurring at any other time during the study. Any AEs and remedial action required will be recorded in the subject's source data. Subjects experiencing AEs will be followed clinically until their health has returned to baseline status or until all parameters have returned to normal or have otherwise been explained.
Oral body temperature changes | BT measured at screening day, check in day, -1 hour relative to dose, 24 hrs postdose and at day 5 after dosed.
  Oral body temperature in °C (BT) will be measured. All measurements will be taken as single readings. Measurements will be repeated once if outside the relevant clinical reference ranges. If repeated, the repeat value will be used in the data analysis. Clinical research unit reference ranges will be applied.
12-lead ECG measurements changes | 12-lead ECG will be measured at: screening day; check in day; 0.5, 1, 6, 12 and 24 hous postdose and day 5 after dosed.
  At check-in, 12-lead ECG will be recorded in triplicate in the supine position for baseline measurements. The average value for each ECG parameter will be calculated as the baseline value. At all other times, a single 12-lead resting ECG with a 10-second rhythm strip will be recorded after the subject has been supine for at least 5 minutes.The 12-lead ECG will be repeated once if either of the following criteria apply:The QTcF is >450 ms; The QTcF change from baseline (check-in) is >60 ms. Additional 12-lead ECGs will be performed at other times if judged to be clinically appropriate or if the ongoing review of the data suggests a more detailed assessment of ECGs is required. The ECG machine will compute the PR, QT and QTc intervals, QRS duration and heart rate. The QT interval will be corrected for heart rate using Fridericia's formula.
Changes in cardiac rhythm monitored by telemetry | Continuous telemetry monitoring from -1 hour to 24 hour relative to dose. Telemetry strips will be printed out at 2, 3, 4 and 5 hours postdose.
  Cardiac rhythm will be monitored by telemetry. Telemetry strips will be printed out at the times indicated in the Study Plan. In addition, staff members will be instructed to print out ECGs if either of the following criteria apply: The QTcF is >450 ms; The QTcF change from baseline (check-in) is >60 ms. In such an event, ECGs will continue to be printed out every 20 minutes until the QTcF value has returned to normal.
Changes in clinical laboratory evaluations | Clinical laboratories evaluations will be measured at: screening day; check in day; -1 hour and 24 hour relative to dose and day 5 after dosed.
  Blood and urine samples will be collected for clinical laboratory evaluations at the times indicated in the Study Plan. Additional clinical laboratory evaluations will be performed at other times if judged to be clinically appropriate or if the ongoing review of the data suggests a more detailed assessment of clinical laboratory safety is required. The following evaluations will be performed: Serum biochemistry, hematology, coagulation, urinalysis and serology.
Changes in blood glucose and phosphorous evaluations | The evaluations will be measured 30 minutes and 1 hour post adminitration of the drug.
  Blood samples will be collected for serum glucose (mg/dL) and phosphorous (mg/dL) evaluations.
Physical examination changes | Physical examination will be performed at: check in day, 1 and 24 hours after dose administration and at day 5 after dosed.
  A full physical examination will be performed at the times indicated in the Study Plan and an abbreviated physical examination may be performed at other times.
Changes in the general wellbeing of the subject | The questionnaire will be conducted every hour for 12 hours postdose and at approximately 24 hours postdose.
  Subjects will be asked to complete a clinical study questionnaire to assess tolerance to the study drug, with the assistance of a suitably trained CRU staff member. Subjects will be asked questions about their general wellbeing and the injection site over the period either since dosing or since the last questionnaire, as applicable. In addition, the injection site will be assessed by the CRU staff member conducting the questionnaire.
Blood pressure changes | BP: measured at screening day, check in day, continuous monitoring during dose day (until 24 hrs) and day 5 after dosed.
  Systolic and Diastolic blood pressure in mmHg (BP), will be measured. At check-in, blood pressure, will be measured in triplicate within a 10-minute window. The median value for systolic and diastolic blood pressure, will be used as the baseline value in the data analysis. All other measurements will be taken as single readings. Measurements will be repeated once if outside the relevant clinical reference ranges. If repeated, the repeat value will be used in the data analysis. Clinical research unit reference ranges will be applied.
Heart rate changes | HR: measured at screening day, check in day, continuous monitoring during dose day (until 24 hrs) and day 5 after dosed.
  Heart rate in bpm (HR) will be measured. At check-in, heart rate will be measured in triplicate within a 10-minute window. The median value for heart rate will be used as the baseline value in the data analysis. All other measurements will be taken as single readings. Measurements will be repeated once if outside the relevant clinical reference ranges. If repeated, the repeat value will be used in the data analysis. Clinical research unit reference ranges will be applied.
Respiratory rate changes | RR: measured at screening day, check in day, continuous monitoring during dose day (until 24 hrs) and day 5 after dosed.
  Respiratory rate in breaths/min (RR) will be measured. At check-in, respiratory rate will be measured in triplicate within a 10-minute window. The median value for respiratory rate will be used as the baseline value in the data analysis. All other measurements will be taken as single readings. Measurements will be repeated once if outside the relevant clinical reference ranges. If repeated, the repeat value will be used in the data analysis. Clinical research unit reference ranges will be applied.
Oxygen saturation changes | OS: measured at screening day, check in day, continuous monitoring during dose day (until 24 hrs) and day 5 after dosed.
  Oxygen saturation in % (OS) will be measured. All measurements will be taken as single readings. Measurements will be repeated once if outside the relevant clinical reference ranges. If repeated, the repeat value will be used in the data analysis. Clinical research unit reference ranges will be applied.

SECONDARY OUTCOMES:
Pharmacokinetic of NAVX-010: Area under the curve from time 0 up to the time of last quantifiable (AUC0-t) plasma concentration. | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the AUC0-t of GTX 2 and GTX 3. The Area under the concentration-time curve from time 0 up to the time of last quantifiable plasma concentration (tlast), calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations.
Pharmacokinetic of NAVX-010: Area under the curve from time 0 to 24 hours postdose (AUC0-24) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the AUC0-24 of GTX 2 and GTX 3. The Area under the concentration-time curve from time 0 to 24 hours postdose, calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations.
Pharmacokinetic of NAVX-010: Area under the curve from time 0 extrapolated to infinity (AUC0-oo) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the AUC0-oo of GTX 2 and GTX 3. The Area under the concentration-time curve from time 0 extrapolated to infinity:
  AUC0-oo= AUC0-t + Clast/λz Where Clast is the last measurable plasma concentration and λz is the terminal elimination rate constant.
Pharmacokinetic of NAVX-010: Percentage of area under the curve that is due to extrapolation from last quantifiable concentration to infinity (%AUCextrap) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the %AUCextrap of GTX 2 and GTX 3. The Percentage of area under the concentration-time curve that is due to extrapolation from last quantifiable concentration to infinity.
Pharmacokinetic of NAVX-010: Maximum observed plasma concentration (Cmax) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the Cmax of GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Time of the maximum observed plasma concentration (tmax) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the tmax of GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Time of last quantifiable plasma concentration (tlast) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the tlast of GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Time before the start of absorption (tlag) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the tlag of GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Apparent plasma terminal elimination half-life (t½) | Plasma samples: pre-dose and 5, 10, 20, 30, and 45 minutes plus 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose.
  Blood samples (approximately 1 x 10 mL) will be taken by venipuncture or cannulation at the times indicated in the Study Plan to calculate the t½ of GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Apparent total plasma clearance (CL/F) | Urine samples evaluation were collected from point of dosing to 12 hours postdose, and from 12 hours to 24 hours postdose.
  Urine will be collected into standard-weight polyethylene containers over the time intervals indicated in the Study Plan. During each collection period, the containers will be stored in a refrigerator at 2 to 8°C. The weight (g) of each collection will be recorded prior to removal of 2 sub-samples (each approximately 4 mL) into suitably labeled polypropylene containers, which will be stored within 4 hours of the end of the collection, at approximately -80°C. The remaining urine will be discarded. A nominal value for specific gravity of 1.018 will be used to calculate urine volume. The CL/F is calculated for GTX 2 and GTX 3 as dose/AUC0-oo.
Pharmacokinetic of NAVX-010: Apparent volume of distribution during the terminal elimination phase (Vz/F) | Urine samples evaluation were collected from point of dosing to 12 hours postdose, and from 12 hours to 24 hours postdose.
  will be stored in a refrigerator at 2 to 8°C. The weight (g) of each collection will be recorded prior to removal of 2 sub-samples (each approximately 4 mL) into suitably labeled polypropylene containers, which will be stored within 4 hours of the end of the collection, at approximately -80°C. The remaining urine will be discarded. A nominal value for specific gravity of 1.018 will be used to calculate urine volume. The Vz/F is calculated for GTX 2 and GTX 3 as CL/λz.
Pharmacokinetic of NAVX-010: Amount of drug excreted in urine (Ae) | Urine samples evaluation were collected from point of dosing to 12 hours postdose, and from 12 hours to 24 hours postdose.
  will be stored in a refrigerator at 2 to 8°C. The weight (g) of each collection will be recorded prior to removal of 2 sub-samples (each approximately 4 mL) into suitably labeled polypropylene containers, which will be stored within 4 hours of the end of the collection, at approximately -80°C. The remaining urine will be discarded. A nominal value for specific gravity of 1.018 will be used to calculate urine volume. The Ae is calculated for GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Percentage of dose excreted in urine (Fe) | Urine samples evaluation were collected from point of dosing to 12 hours postdose, and from 12 hours to 24 hours postdose.
  will be stored in a refrigerator at 2 to 8°C. The weight (g) of each collection will be recorded prior to removal of 2 sub-samples (each approximately 4 mL) into suitably labeled polypropylene containers, which will be stored within 4 hours of the end of the collection, at approximately -80°C. The remaining urine will be discarded. A nominal value for specific gravity of 1.018 will be used to calculate urine volume. The Fe is calculated for GTX 2 and GTX 3.
Pharmacokinetic of NAVX-010: Renal clearance (CLR) | Urine samples evaluation were collected from point of dosing to 12 hours postdose, and from 12 hours to 24 hours postdose.
  will be stored in a refrigerator at 2 to 8°C. The weight (g) of each collection will be recorded prior to removal of 2 sub-samples (each approximately 4 mL) into suitably labeled polypropylene containers, which will be stored within 4 hours of the end of the collection, at approximately -80°C. The remaining urine will be discarded. A nominal value for specific gravity of 1.018 will be used to calculate urine volume. The CLR is calculated for GTX 2 and GTX 3.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Whitehurst, MD, Principal Investigator — Covance Clinical Research Unit, Evansville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Food and Drug Administration Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. — http://www.fda.gov/downloads/Drugs/Guidance/UCM078932.pdf